CLINICAL TRIAL: NCT05474482
Title: Comparison of Kinesio Taping With and Without Combined Exercise Program on Pain and Quality of Life in Primary Dysmenorrhea
Brief Title: Kinesio Taping With and Without Exercise Program in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0513
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea, Kinesiology taping, Menstruation
MeSH Terms: conditions — Dysmenorrhea | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- kinesio taping with 75 to 100 % stretch and exercises (Experimental): Kinesio taping with stretching exercises and yoga will be given to patients for 8 weeks.
  Interventions: Other: kinesio taping with exercises
- kinesio taping without exercises (Experimental): Kinesio taping alone will be given to patients for 8 weeks.
  Interventions: Other: Kinesio taping without exercises
- kinesio taping without stretch to tape (Active Comparator): kinesio taping without any stretch, applied as control for 8 weeks.
  Interventions: Other: Kinesio taping without stretch as control

INTERVENTIONS:
Other: kinesio taping with exercises — Kinesio taping with full stretch of 75 to 100 % for 2 days session per week and exercises for 3 days session per week for total 8 weeks.
  Arms: kinesio taping with 75 to 100 % stretch and exercises
Other: Kinesio taping without exercises — Kinesio taping with a full stretch of 75 to 100 % for 2 days session per week without exercises for 8 weeks.
  Arms: kinesio taping without exercises
Other: Kinesio taping without stretch as control — kinesio taping without any stretch for 2 days session per week for total 8 weeks.
  Arms: kinesio taping without stretch to tape

SUMMARY:
Primary dysmenorrhea (PD) is a common gynecological problem among adolescents and adult women. Treatment of PD includes various drugs and therapies such as kinesio taping (KT) and exercise. There are various studies that have individually explored the effects of KT and combined exercises. A randomized controlled trial (RCT) will be conducted to compare the effects of KT combined a combined exercise program and the effects of KT alone on pain and quality of life in females suffering from PD.

DETAILED DESCRIPTION:
Primary dysmenorrhea (PD) is a common gynecological problem among adolescents and adult women. Treatment of PD includes various drugs and therapies such as kinesio taping (KT) and exercise. There are various studies that have individually explored the effects of KT and combined exercises. A randomized controlled trial (RCT) will be conducted to compare the effects of KT combined a combined exercise program and the effects of KT alone on pain and quality of life in females suffering from PD. The study will involve 45 women who experience dysmenorrhea. divided into three groups, group A, group B and Group C. Group A will receive the combined exercise program (The exercise protocol which included stretching exercises, yoga position, Kegel exercise, bridging exercise) for 45 minutes with 3 sessions per week for eight weeks. The Group A will receive KT intervention for two days per week from the estimated day of ovulation till the next period occurs, for eight weeks. The group B will receive KT that is used to treat the symptoms of primary dysmenorrhea for 45 minutes with 2 sessions per week for eight weeks. The Group C will receive conventional therapy with 3 sessions per week to eight weeks. Numeric pain rating scale (NPRS), Short form 36 Questionnaire (SF-36) and Menstrual symptom questionnaire (MSQ) will be used to assess the pain and quality of life at baseline and at the end of 8th week.Total duration of study will be six months. Physiotherapy can be a very successful treatment for PD with the benefit that the patient may occasionally be able to carry out the treatment independently. recommendations for manual therapy, acupressure, Kinesio tape, electrotherapy, and other forms of treatment. There have also been discussions about therapeutic activities or progressive relaxation techniques.

It is stated in literature that most effective exercise programs were stretching and isometric exercises for 8 weeks for pain intensity and duration, yoga for 12 weeks for pain intensity and quality of life, and aerobic exercises for 12 weeks for quality of life and KT for 12 weeks for pain and quality of life in PD. There are many various tapes available, each with a different type, substance, and application, according to the most recent research in 2021.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 30 who are nulliparous and have normal menstrual cycles (28 to 7 days).
* Menstrual pain severity rated at 4 or higher on the NPRS over the previous six months.

Exclusion Criteria:

* Secondary dysmenorrhea Pelvic surgery (rectum and anal problems, etc.), pelvic organ prolapses, and malignant conditions (uterine cancer, ovarian cancer, cervical cancer, etc.)
* Utilizing oral contraceptives for at least six months before.
* Allergic to KT tape
* Use of antidepressants

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
MSQ | 6 months
  Menstrual symptoms were assessed using the Menstrual Symptom Questionnaire (MSQ). The questionnaire has 24 items; 19 of them (emotional, physical, and pain) assess symptoms, and three examine symptom management strategies. The following is how the things are rated using a Likert-style scale: 1 denotes never, 2 rare, 3 irregular, 4 often, and 5 constant.

SECONDARY OUTCOMES:
SF36 | 6 months
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study
NPRS | 6 months
  NPRS with each centimetre denoting one unit of pain severity, to indicate how much pain they were experiencing. "0" meant there was no pain, while "10" meant there was a lot of agonyas used to measure pain. The participants marked a "x" on a 10 cm line,

CONTACTS AND LOCATIONS:
Overall Officials: Afifa Safdar, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Johar Institute of Professional Studies nabi bakhsh stop, lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toprak Celenay S, Kavalci B, Karakus A, Alkan A. Effects of kinesio tape application on pain, anxiety, and menstrual complaints in women with primary dysmenorrhea: A randomized sham-controlled trial. Complement Ther Clin Pract. 2020 May;39:101148. doi: 10.1016/j.ctcp.2020.101148. Epub 2020 Mar 18. PMID 32379680
- [Background] Kirmizigil B, Demiralp C. Effectiveness of functional exercises on pain and sleep quality in patients with primary dysmenorrhea: a randomized clinical trial. Arch Gynecol Obstet. 2020 Jul;302(1):153-163. doi: 10.1007/s00404-020-05579-2. Epub 2020 May 15. PMID 32415471
- [Background] Mejias-Gil E, Garrido-Ardila EM, Montanero-Fernandez J, Jimenez-Palomares M, Rodriguez-Mansilla J, Gonzalez Lopez-Arza MV. Kinesio Taping vs. Auricular Acupressure for the Personalised Treatment of Primary Dysmenorrhoea: A Pilot Randomized Controlled Trial. J Pers Med. 2021 Aug 19;11(8):809. doi: 10.3390/jpm11080809. PMID 34442453
- [Background] Lopez-Liria R, Torres-Alamo L, Vega-Ramirez FA, Garcia-Luengo AV, Aguilar-Parra JM, Trigueros-Ramos R, Rocamora-Perez P. Efficacy of Physiotherapy Treatment in Primary Dysmenorrhea: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jul 23;18(15):7832. doi: 10.3390/ijerph18157832. PMID 34360122
- [Background] Blakey H, Chisholm C, Dear F, Harris B, Hartwell R, Daley AJ, Jolly K. Is exercise associated with primary dysmenorrhoea in young women? BJOG. 2010 Jan;117(2):222-4. doi: 10.1111/j.1471-0528.2009.02220.x. PMID 19459861
- [Background] Tomas-Rodriguez MI, Palazon-Bru A, Martinez-St John DRJ, Toledo-Marhuenda JV, Asensio-Garcia MDR, Gil-Guillen VF. Effectiveness of medical taping concept in primary dysmenorrhoea: a two-armed randomized trial. Sci Rep. 2015 Nov 13;5:16671. doi: 10.1038/srep16671. PMID 26564807
- [Background] Dogan H, Eroglu S, Akbayrak T. The effect of kinesio taping and lifestyle changes on pain, body awareness and quality of life in primary dysmenorrhea. Complement Ther Clin Pract. 2020 May;39:101120. doi: 10.1016/j.ctcp.2020.101120. Epub 2020 Feb 22. PMID 32379659